CLINICAL TRIAL: NCT02246881
Title: An Open Study to Compare the Pharmacokinetics and Safety of Current Factor VIII Concentrate and Optivate® in Severe Haemophilia A Patients.
Brief Title: A Study to Compare the Pharmacokinetics and Safety of Current Factor VIII Concentrate and Optivate® in Haemophilia A.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 8VWFPK
Record Dates: First submitted 2014-09-02; First posted 2014-09-23 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases | interventions — optivate; Factor VIII

ARMS (2):
- Current Factor VIII (Active Comparator): Optivate® (Human Coagulation Factor VIII)
  Interventions: Biological: Optivate® (Human Coagulation Factor VIII)
- Optivate® (Experimental): Optivate® (Human Coagulation Factor VIII)
  Interventions: Biological: Optivate® (Human Coagulation Factor VIII)

INTERVENTIONS:
Biological: Optivate® (Human Coagulation Factor VIII)

SUMMARY:
The main objective of the study is to compare the pharmacokinetics of Optivate® with the subject's current FVIII concentrate when given as a bolus dose of 50IU/kg. The secondary objective is to compare the first and second pharmacokinetic assessments on Optivate® (and recovery if a subject changes batch) to evaluate Optivate® in terms of clinical tolerance and safety.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated subjects with severe Haemophilia A (<2% basal FVIII activity) without inhibitor to Factor VIII, at least 12 years of age, currently receiving FVIII concentrate and with more than 20 exposure days.

Exclusion Criteria:

-

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-10; Primary Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
PK parameters for FVIII:C | Pre-dose, 15, 30 min, 1, 3, 6, 9, 24, 28, 32, 48 hours post-dose

CONTACTS AND LOCATIONS:
Locations (8):
- Poland (3):
  - Klinika Haematologii, Akademia Medyczna w Gdansku, ul., Debinki 7, 80-211 Gdansk
  - Klinika Haematologii, Akademia Medyczna w Lublinie, ul., Dr K Jaczewskiego 8, 20-090, Lublin
  - Klinika Haematologii, Akademia Medyczna w Lodzi, ul., Pabianicka 62, 93-513 Lodz
- United Kingdom (5):
  - Haemophilia Centre, Addenbrooke's Hospital, Hills Road, Cambridge, Cambridgeshire
  - Haemophilia Centre, University Hospital, Queens Medical Centre, Clifton Boulevard, Nottingham
  - Sheffield Haemophilia & Thrombosis Centre, Royal Hallamshire Hospital, Glossop Road, Sheffield
  - Haemophilia Centre, University Dept. of Haemophilia, Manchester Royal Infirmary, Manchester
  - Haemophilia Centre, Southampton General Hospital, Tremona Road, Southampton

REFERENCES:
- See also: Related Info — http://www.bpl.co.uk